CLINICAL TRIAL: NCT03023566
Title: Intra-individual Open-label, Single Center Study to Compare Unenhanced MRI With Dotarem Enhanced MRI in Pediatric and Neonatal Patient Population (<18years)
Brief Title: Intra-individual Open-label, Single Center Study to Compare Unenhanced MRI With Dotarem Enhanced MRI
Status: Completed | Type: Observational
Sponsor: Phoenix Children's Hospital (Other)
Collaborators: Guerbet (Industry)
Responsible Party: Principal Investigator, Jeffrey Miller, MD, Staff Physician, Vice Chair of Radiology, Phoenix Children's Hospital
Other Study IDs: PCH IRB#16-102
Record Dates: First submitted 2017-01-12; First posted 2017-01-18 (Estimated); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Brain Diseases
Keywords: Dotarem; MRI; pediatric; safety; efficacy
MeSH Terms: conditions — Brain Diseases | interventions — gadoterate meglumine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

GROUPS / COHORTS (1):
- Dotarem Enhanced MRI: All pediatric patients (< 18 years) scheduled for clinically indicated contrast enhanced MRI (Brain MRI with/without contrast) will receive a single IV bolus injection of Dotarem at a dose of 0.1 mmol/kg bw at a flow rate of 1-2 mL/sec followed by saline flush (routine/ standard of care).
  Interventions: Drug: Dotarem

INTERVENTIONS:
Drug: Dotarem — Dotarem at dose of 0.1 mmol/kg of body weight (routine/standard of care)
  Other Names: gadoterate meglumine

SUMMARY:
The goal of this study is to evaluate safety and efficacy of Dotarem enhanced MRI in pediatric and neonatal population who are referred for contrast enhanced MRI at Phoenix Children's Hospital.

DETAILED DESCRIPTION:
Phoenix Children's Hospital (PCH) performs approximately 200 contrast enhanced MRI procedures per month. Recently PCH changed its MRI contrast agent from the linear contrast agent Magnevist to the macrocyclic contrast agent Dotarem. The goal of this study is to evaluate safety and efficacy of Dotarem enhanced MRI in pediatric and neonatal population who are referred for contrast enhanced MRI at PCH.

The study is designed as a single center, open label comparison of unenhanced MRI with Dotarem enhanced MRI in pediatric patient population (<18years). The comparison will be performed intra-individually by 3 independent blinded radiologists. Overall, the study population will consist of 250 pediatric patients who are indicated for contrast enhanced MRI. The safety follow-up period will be 24 (+/- 4) hours post injection of Dotarem and includes the assessment of physical examinations and vital signs as well as the assessment of AEs.

ELIGIBILITY:
Inclusion Criteria:

* Any patient under 18 years of age who is scheduled for contrast enhanced MRI examination as part of their standard of care.
* Patients who are willing to undergo contrast enhanced MRI procedure
* Patients who are willing to comply with the study procedures (e.g. being followed-up for 24 hours after MRI procedure).
* Patients who have given their fully informed and written consent voluntarily.

Exclusion Criteria:

* Patients receiving an MRI exam without contrast.
* Patients who are pregnant, lactating or who are > 11 years old and have not had a negative urine pregnancy test the same day as administration of Dotarem. The manufacturer's instructions for performing the urinary pregnancy test are to be followed.
* Having an underlying disease or concomitant medication which may interfere with efficacy or safety evaluations as planned in this study.
* Patients with a Glomerular Filtration Rate (GFR) < 30.
* Having received any investigational drug within 30 days prior to entering this study or who are planned to receive any investigational drug during the 24 (+ / - 4) hour safety follow-up period.
* Not being able to remain lying down for at least 45 - 60 min (e.g. patients with unstable angina, dyspnea at rest, severe pain at rest, severe back pain).
* Presenting with history of anaphylactoid or anaphylactic reaction to any allergen including drugs and contrast agents .
* Patients who have received any other contrast medium within 24 hours prior to Dotarem injection or are scheduled to receive any other contrast medium within the follow-up period.
* Being clinically unstable and whose clinical course during the 24 (+ / - 4) hours observation period is unpredictable.
* Being scheduled for, or likely to require, any surgical intervention within 24 hours before or within the follow-up period.
* Having any contraindication to MRI examination (e.g. pacemaker, recent wound clips, and severe claustrophobia).
* Having been previously enrolled in this study.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will consist of N = 250 pediatric patients (< 18 years) who are indicated for contrast enhanced MRI.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2017-11-12 (Actual); Study Completion 2017-11-12 (Actual)

PRIMARY OUTCOMES:
Overall lesion visualization and characterization | 24 - 48 hours
  Overall lesion visualization and characterization, based on assessment of (1) lesion border delineation, (2) internal morphology and (3) degree of contrast enhancement. All images from "Pre" (unenhanced MRI) and "Paired" (unenhanced + enhanced) MRI will be evaluated independently by the 3 independent readers and are rated on a 3-point scale as unevaluable (0), seen but imperfectly (1) or seen completely/perfectly (2). The primary statistical analysis compared unenhanced MRI to combined MRI. The efficacy of Dotarem is expected to be demonstrated for at least 2 out of 3 readers independently meeting a statistically significant positive difference between the mean "Paired" score and the mean "Pre" score at patient level for each co primary endpoints.

SECONDARY OUTCOMES:
Efficacy of enhanced MRI compared to unenhanced MRI | 24 - 48 hours
  Efficacy of enhanced MRI compared to unenhanced MRI, based on (1) lesion counting, (2) signal intensity measurements, (3) image quality evaluation, and (4) diagnostic confidence (defined on 1-5 scale; 1= no confidence and 5 represents very high confidence
Assessment of adverse events (AEs) | 24 hours (+ / - 4 hours)
  Assessment of adverse events (AEs), volunteered, observed or elicited by vital signs, physical examination, and continuous monitoring of AEs from the beginning of Dotarem injection until end of the follow-up period of 24 (+ / - 4) hours after contrast administration.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey H Miller, MD, Principal Investigator — Phoenix Children's Hospital
Locations (1):
- Phoenix Children's Hospital, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No